CLINICAL TRIAL: NCT04747860
Title: Generalization of Fear of Movement-related Pain and Avoidance Behavior as Predictors of Work Resumption After Back Surgery. A Prospective Study
Brief Title: Predictors of Work Resumption After Back Surgery
Acronym: WABS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: RIZIV (Unknown)
Responsible Party: Principal Investigator, Johan Vlaeyen, Principal Investigator, Professor, KU Leuven
Other Study IDs: S63018; ctu2019088 (Registry Identifier: FearedBack ZOL); AZGS2020051 (Registry Identifier: FearedBack AZ Groeninge)
Record Dates: First submitted 2018-08-20; First posted 2021-02-10 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Low Back Pain
Keywords: Low back pain; Back surgery; Postoperative pain; Predictors of return to work; Fear of movement-related pain; Avoidance; Fear generalization; Avoidance generalization; Disability; Quality of life
MeSH Terms: conditions — Low Back Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, longitudinal study aims to identify modifiable predictors of return to work after back surgery.

DETAILED DESCRIPTION:
Background | Over the past decade, the number of back surgeries in Belgium has substantially increased. However, even after an anatomically successful surgery, 10% to 40% of the patients continue to report pain complaints, causing personal suffering and an enormous economic burden. The specific factors that can predict individual trajectories in postoperative pain, recovery, and work resumption are currently largely unknown.

Aim | The aim of this study is to identify modifiable predictors of work resumption after back surgery.

Methods | In this multisite, prospective, longitudinal study, 300 individuals undergoing back surgery will be followed one-year post-surgery. Prior to surgery, the participants will perform a behavioral computer task to assess fear of movement-related pain and avoidance behavior, and their generalization. In addition, participants will complete questionnaires to assess preoperative fear of movement-related pain, avoidance behavior, optimism, expectancies towards recovery and work resumption, and the duration and severity of the pain before the surgery. Immediately after surgery, as well as six weeks, three months, six months, and twelve months postoperatively, sustainable work resumption, pain severity, disability, and quality of life will be assessed.

Hypothesis | The primary hypothesis is that generalization of fear of movement-related pain and avoidance behavior will negatively affect sustainable work resumption after back surgery. Second, the investigators hypothesize that generalization of fear of movement-related pain and avoidance behavior, negative expectancies towards recovery and work resumption, longer pain duration, and more severe pain before the surgery will negatively affect work resumption, pain severity, disability, and quality of life after back surgery. In contrast, positive expectancies towards recovery and work resumption and optimism are expected positively influence work resumption, pain severity, disability, and quality of life.

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 55 years
* Proper mastery of the Dutch, English and/or French language
* Intermittent or constant invalidating lumbosciatica for less than 1 year prior to the planned surgery
* Discogenic or stenotic radicular pain in the leg(s) that will be treated surgically by performing a decompression without it leading to fusion and/or fixation
* Self-employed or has an employment contract, and is on sick leave for less than 1 year at the day of the surgery

Exclusion criteria:

* Treated (ambulant or residential) for substance abuse, suicidal ideation or a psychotic disorder in the year before the consult with the surgeon. Ty
* At least one back surgery in the last 5 years
* Presence of a comorbid condition (e.g. a severe neurological deficit, a pulmonary embolism, permanent paralysis, and another pain problem in the limbs), which may affect the pain, the outcome of the surgery, the duration of the rehabilitation, and/or the patient's capacity to return to work during the course of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with low back pain who will undergo back surgery
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported (sustainable) work resumption assessed by self-report questionnaires | 6 weeks post-surgery
  The investigators make a distinction between being fit for work, work resumption, and sustainable work resumption. Being fit for work will be operationalized by not receiving disability benefits. Work resumption will be operationalized by being at work without receiving disability benefits, and time to relapse. Time to relapse is defined as the time for participants to be in sick leave again after being fit for work. Sustainable work resumption will be operationalized by being at work for at least three consecutive months without receiving disability benefits. In addition, the duration of work resumption will be measured.
Self-reported (sustainable) work resumption assessed by self-report questionnaires | 3 months post-surgery
  The investigators make a distinction between being fit for work, work resumption, and sustainable work resumption. Being fit for work will be operationalized by not receiving disability benefits. Work resumption will be operationalized by being at work without receiving disability benefits, and time to relapse. Time to relapse is defined as the time for participants to be in sick leave again after being fit for work. Sustainable work resumption will be operationalized by being at work for at least three consecutive months without receiving disability benefits. In addition, the duration of work resumption will be measured.
Self-reported (sustainable) work resumption assessed by self-report questionnaires | 6 months post-surgery
  The investigators make a distinction between being fit for work, work resumption, and sustainable work resumption. Being fit for work will be operationalized by not receiving disability benefits. Work resumption will be operationalized by being at work without receiving disability benefits, and time to relapse. Time to relapse is defined as the time for participants to be in sick leave again after being fit for work. Sustainable work resumption will be operationalized by being at work for at least three consecutive months without receiving disability benefits. In addition, the duration of work resumption will be measured.
Self-reported (sustainable) work resumption assessed by self-report questionnaires | 12 months post-surgery
  The investigators make a distinction between being fit for work, work resumption, and sustainable work resumption. Being fit for work will be operationalized by not receiving disability benefits. Work resumption will be operationalized by being at work without receiving disability benefits, and time to relapse. Time to relapse is defined as the time for participants to be in sick leave again after being fit for work. Sustainable work resumption will be operationalized by being at work for at least three consecutive months without receiving disability benefits. In addition, the duration of work resumption will be measured.

SECONDARY OUTCOMES:
Self-reported ratings of how much pain the participants experiences, assessed by one question of the short Örebro Musculoskeletal Pain Screening Questionnaire (ÖMPSQ) | 6 weeks post-surgery
  Pain severity will be operationalized as the intensity of the pain, and will be assessed by one questions of the short ÖMPSQ (Linton et al., 2011). Participants are requested to answer this item (i.e., How would you rate the pain that you have had during the past week?) on a numerical rating scale with labels from 0 = no pain to 10 = pain as bad as it could be. The score on this item will be used as a measure of pain severity before and immediately after the surgery (as baseline measures) and six weeks, three months, six months and twelve months post-surgery.
Self-reported ratings of how much pain the participants experiences, assessed by one question of the short ÖMPSQ | 3 months post-surgery
  Pain severity will be operationalized as the intensity of the pain, and will be assessed by one questions of the short ÖMPSQ (Linton et al., 2011). Participants are requested to answer this item (i.e., How would you rate the pain that you have had during the past week?) on a numerical rating scale with labels from 0 = no pain to 10 = pain as bad as it could be. The score on this item will be used as a measure of pain severity before and immediately after the surgery (as baseline measures) and six weeks, three months, six months and twelve months post-surgery.
Self-reported ratings of how much pain the participants experiences, assessed by one question of the short ÖMPSQ | 6 months post-surgery
  Pain severity will be operationalized as the intensity of the pain, and will be assessed by one questions of the short ÖMPSQ (Linton et al., 2011). Participants are requested to answer this item (i.e., How would you rate the pain that you have had during the past week?) on a numerical rating scale with labels from 0 = no pain to 10 = pain as bad as it could be. The score on this item will be used as a measure of pain severity before and immediately after the surgery (as baseline measures) and six weeks, three months, six months and twelve months post-surgery.
Self-reported ratings of how much pain the participants experiences, assessed by one question of the short ÖMPSQ | 12 months post-surgery
  Pain severity will be operationalized as the intensity of the pain, and will be assessed by one questions of the short ÖMPSQ (Linton et al., 2011). Participants are requested to answer this item (i.e., How would you rate the pain that you have had during the past week?) on a numerical rating scale with labels from 0 = no pain to 10 = pain as bad as it could be. The score on this item will be used as a measure of pain severity before and immediately after the surgery (as baseline measures) and six weeks, three months, six months and twelve months post-surgery.
Self-reported ratings of the extent that pain interferes with functioning, assessed by Pain Disability Index (PDI) | 6 weeks post-surgery
  Disability will be operationalized as the degree to which pain interferes with functioning, and will be assessed by the Pain Disability Index (PDI) questionnaire (Pollard, 1984). The PDI is a self-report questionnaire that measures the degree to which pain interferes with functioning in seven areas: i.e., family/home responsibilities, recreation, social activity, occupation, sexual behavior, self-care, and life-support activity (Tait et al., 1990). Ratings for each item range from 0 = no disability to 5 = total disability. A total score will be calculated as a reliable and valid (Tait et al., 1990) measure of degree of disability before and immediately after the surgery (as baseline measures) and six weeks, three months, six months and twelve months post-surgery.
Self-reported ratings of the extent that pain interferes with functioning, assessed by Pain Disability Index (PDI) | 3 months post-surgery
  Disability will be operationalized as the degree to which pain interferes with functioning, and will be assessed by the Pain Disability Index (PDI) questionnaire (Pollard, 1984). The PDI is a self-report questionnaire that measures the degree to which pain interferes with functioning in seven areas: i.e., family/home responsibilities, recreation, social activity, occupation, sexual behavior, self-care, and life-support activity (Tait et al., 1990). Ratings for each item range from 0 = no disability to 5 = total disability. A total score will be calculated as a reliable and valid (Tait et al., 1990) measure of degree of disability before and immediately after the surgery (as baseline measures) and six weeks, three months, six months and twelve months post-surgery.
Self-reported ratings of the extent that pain interferes with functioning, assessed by Pain Disability Index (PDI) | 6 months post-surgery
  Disability will be operationalized as the degree to which pain interferes with functioning, and will be assessed by the Pain Disability Index (PDI) questionnaire (Pollard, 1984). The PDI is a self-report questionnaire that measures the degree to which pain interferes with functioning in seven areas: i.e., family/home responsibilities, recreation, social activity, occupation, sexual behavior, self-care, and life-support activity (Tait et al., 1990). Ratings for each item range from 0 = no disability to 5 = total disability. A total score will be calculated as a reliable and valid (Tait et al., 1990) measure of degree of disability before and immediately after the surgery (as baseline measures) and six weeks, three months, six months and twelve months post-surgery.
Self-reported ratings of the extent that pain interferes with functioning, assessed by Pain Disability Index (PDI) | 12 months post-surgery
  Disability will be operationalized as the degree to which pain interferes with functioning, and will be assessed by the Pain Disability Index (PDI) questionnaire (Pollard, 1984). The PDI is a self-report questionnaire that measures the degree to which pain interferes with functioning in seven areas: i.e., family/home responsibilities, recreation, social activity, occupation, sexual behavior, self-care, and life-support activity (Tait et al., 1990). Ratings for each item range from 0 = no disability to 5 = total disability. A total score will be calculated as a reliable and valid (Tait et al., 1990) measure of degree of disability before and immediately after the surgery (as baseline measures) and six weeks, three months, six months and twelve months post-surgery.
Self-reported ratings of how satisfied the participants is with his/her life overall, assessed by one item of the Riverside Life Satisfaction Scale | 6 weeks post-surgery
  Quality of life will be operationalized as satisfaction with life. It will be measured by the one item of the Riverside Life Satisfaction Scale (RLSS) with the highest factor loading (Margolis et al., 2019). Participants are requested to answer this item (i.e., I am satisfied with my life overall.) on a 7-point Likert scale ranging from strongly disagree to strongly agree.
Self-reported ratings of how satisfied the participants is with his/her life overall, assessed by one item of the Riverside Life Satisfaction Scale | 3 months post-surgery
  Quality of life will be operationalized as satisfaction with life. It will be measured by the one item of the Riverside Life Satisfaction Scale (RLSS) with the highest factor loading (Margolis et al., 2019). Participants are requested to answer this item (i.e., I am satisfied with my life overall.) on a 7-point Likert scale ranging from strongly disagree to strongly agree.
Self-reported ratings of how satisfied the participants is with his/her life overall, assessed by one item of the Riverside Life Satisfaction Scale | 6 months post-surgery
  Quality of life will be operationalized as satisfaction with life. It will be measured by the one item of the Riverside Life Satisfaction Scale (RLSS) with the highest factor loading (Margolis et al., 2019). Participants are requested to answer this item (i.e., I am satisfied with my life overall.) on a 7-point Likert scale ranging from strongly disagree to strongly agree.
Self-reported ratings of how satisfied the participants is with his/her life overall, assessed by one item of the Riverside Life Satisfaction Scale | 12 months post-surgery
  Quality of life will be operationalized as satisfaction with life. It will be measured by the one item of the Riverside Life Satisfaction Scale (RLSS) with the highest factor loading (Margolis et al., 2019). Participants are requested to answer this item (i.e., I am satisfied with my life overall.) on a 7-point Likert scale ranging from strongly disagree to strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Johan WS Vlaeyen, PhD, Principal Investigator — Health Psychology, KU Leuven
Locations (9):
- Belgium (9):
  - GasthuisZusters Antwerpen (GZA) (campus Sint-Augustinus), department of Neurosurgery, Wilrijk, Antwerpen
  - Centre Hospitalier de Wallonie picarde (CHwapi), department of Neurosurgery, Tournai, Henegouwen
  - Ziekenhuis Oost-Limburg, department of Neurosurgery, Genk, Limburg
  - Mariaziekenhuis Noord-Limburg, departement of Orthopedics, Overpelt, Limburg
  - AZ Sint-Lucas Gent, departement of Orthopedics, Ghent, Oost-Vlaanderen
  - University Hospital Leuven, department of Neurosurgery, Leuven, Vlaams-Brabant
  - Regionaal Ziekenhuis Heilig Hart Tienen, department of Neurosurgery, Tienen, Vlaams-Brabant
  - AZ Groeninge (campus kennedylaan), department of Neurosurgery, Kortrijk, West-Vlaanderen
  - Imeldaziekenhuis, department of Neurosurgery, Bonheiden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masuy R, Bamelis L, Bogaerts K, Depreitere B, De Smedt K, Ceuppens J, Lenaert B, Lonneville S, Peuskens D, Van Lerbeirghe J, Van Schaeybroeck P, Vorlat P, Zijlstra S, Meulders A, Vlaeyen JWS. Generalization of fear of movement-related pain and avoidance behavior as predictors of work resumption after back surgery: a study protocol for a prospective study (WABS). BMC Psychol. 2022 Feb 22;10(1):39. doi: 10.1186/s40359-022-00736-5. PMID 35193697